CLINICAL TRIAL: NCT03272282
Title: Paperless Partograph Evaluation of Labour
Brief Title: Paperless Parotograph in Evaluation of Labour
Acronym: labourRecord
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ayman darder, principal investigator, Assiut University
Other Study IDs: paperlesspartograph
Record Dates: First submitted 2017-08-23; First posted 2017-09-05 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Labor Complication
Keywords: WHO PARTOGRAPG.OBSTRUCTED LABOUR. managment of labour
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — By fellowing women during labour when cervical dilation reach 4cm in active phase of labour all women with inclusion criteria are recorded all women with exclusion criteria are excluded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Using Paperless partograph management of labour as simple tool to prevent obstructed labour or prolonged labour or its complications at the mother or her fetus

DETAILED DESCRIPTION:
WHO PARTOGRAPH is very work load need more time and more stuff in both treaning and learning for plotting and for drowning but inside labour room needing simple partograph playing the simple partograph beast role in management of labour and stand test against time for saving live of labour women and her child Paperless parotograph can help obestitricianes to talk decision about when to transferr the labourus women to higher centers on to make medical intervention or what time to end labour by caesarian section

ELIGIBILITY:
Inclusion Criteria:

* women ln active phase of labour
* With single pregnanncy
* living fetus
* cephalic presentation
* occipt anterior
* 36 weak gestional age up to full term

Exclusion Criteria:

* preterm . .or women with antipartum hemorrhage .
* or multipregnanncy
* previous utrine surgery
* or abnormal cardiotocograph(CTG )PATTERN
* or any heart disease of mother or his fetus

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women ln active phase of labour cerivical dilution 4cm or more
Study Population: By following women during labour using well structured questions developed by researcher and filling well designed Paperless partograph stumped THE collected data will be analysed using special computer program SPSS tactical program for social science
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-09-12 (Estimated); Study Completion 2017-09-12 (Estimated)

PRIMARY OUTCOMES:
Progress of labour | up to 5 months
  Cervical dilatation 1 cm / hour

SECONDARY OUTCOMES:
Charcteristics of new_born | up to 1 month
  Apgar score at1minute and Apgar score at 5minutes
Time taken after ALERT EDT | up to 2 months
  Primgravida and Multipara

OTHER OUTCOMES:
Mode of delivery | up to 9 weeks
  Normal vaginal delivery or caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: mohamed khalaph, Study Director — assiut universty faculity of medicine; ahmad abass, Study Chair — assiut university faclity of meficibe
Locations (2):
- Egypt (2):
  - Faculity of Medicine Assiut University, Asyut, Asyut Governorate
  - Faculity of Medicine, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fatehi F, Gray LC, Wootton R. How to improve your PubMed/MEDLINE searches: 3. advanced searching, MeSH and My NCBI. J Telemed Telecare. 2014 Mar;20(2):102-12. doi: 10.1177/1357633X13519036. PMID 24614997
- [Result] Jadad AR, McQuay HJ. Searching the literature. Be systematic in your searching. BMJ. 1993 Jul 3;307(6895):66. doi: 10.1136/bmj.307.6895.66-a. No abstract available. PMID 8343701
- [Result] Chang AA, Heskett KM, Davidson TM. Searching the literature using medical subject headings versus text word with PubMed. Laryngoscope. 2006 Feb;116(2):336-40. doi: 10.1097/01.mlg.0000195371.72887.a2. PMID 16467730
- See also: more information can present in thishomepage — http://www.iiste.org/journals
- Available data/document: Study Protocol: prospective auther of journals — http://www.iiste.org/journals/ — All the journals articles are amiable online to the reader all over the world without financially legal barriers